CLINICAL TRIAL: NCT02223845
Title: Randomised Controlled Trial of the Effect of Music on Women Undergoing Assisted Reproductive Technology Treatments.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHMO&G0201
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Anxiety
Keywords: Music, Anxiety, IVF
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music (Experimental): Played music during embryo transfer
  Interventions: Other: Music
- Control (No Intervention): No music played during embryo transfer

INTERVENTIONS:
Other: Music — Self-selected music played via headphones
  Arms: Music

SUMMARY:
To investigate whether listening to music at the time of embryo transfer reduces anxiety levels in women undergoing assisted conception treatment.

DETAILED DESCRIPTION:
An assessor-blinded randomized case control study in an IVF center, England UK will randomise women into 'music' (listened to self-selected music during embryo transfer) or 'control' (no music) groups. Participants will complete the Spielberger State-Trait Anxiety Inventory prior to, and immediately following a post-treatment observation period. Total scores will be compared.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were women aged between 25-40 years, undergoing IVF or ICSI with fresh or frozen embryos to completion from February 2013 to December 2013.

Exclusion Criteria:

Women unable to consent or with hearing impairment were excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Anxiety level | 20 minutes
  Participants completed the Spielberger State-Trait Anxiety Inventory prior to, and immediately following a post-treatment observation period. Total scores were compared.

SECONDARY OUTCOMES:
Background anxiety | 20 minutes prior to ET
  Background anxiety is the state anxiety of the women
Quality of life scores | 20 minutes prior to ET
  Quality of life scores as measured by a specific fertility questionnaire
Ongoing pregnancy rate | At 2 weeks and 6 weeks after ET
  Ongoing pregnancy rate as measured by BHG and ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Complete Fertility, Southampton, Hampshire, United Kingdom